CLINICAL TRIAL: NCT06853704
Title: The Clinical Effects of Using Collagen Matrix in Papilla Augmentation: a Prospective Clinical Trial.
Brief Title: The Clinical Effects of Using Collagen Matrix in Papilla Augmentation: a Prospective Clinical Trial. Augmenting Fibro-Gide in Interdental Area Using Tunneling Technique to Treat Black Triangles (Papilla Loss)
Acronym: TPA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JUST university IRBID Jordan
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dental Papilla Loss, Black Triangles; Black Traingles; Interdental Papillae Reconstruction; Interdental Papilla Augmentation; Interdental Papilla Loss
Keywords: papilla; papilla loss; tunnelling; papilla augmentaion

STUDY DESIGN:
Intervention Model Description: it's a clinical trial to see the effects of collagen matrix, using it for the first time in papilla augmentation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): on group of patients with papilla loss
  Interventions: Procedure: papillary unit advancement

INTERVENTIONS:
Procedure: papillary unit advancement — collagen matrix augmentation in papilla area using tunneling technique, up to my knowledge, it's the first time to use collagen matrix in treating papilla, in less invasive approach, only though tunneling with no primary and secondary incisions.
  so, the technique is designed to be less invasive, maximizing papillary blood supply.
  and to use xeno collagen matrix instead of connective tissue graft used in previous study. so ~ less morbidity, less postoperative pain with no Donar graft site .

SUMMARY:
Black triangles, also known as open gingival embrasures, are usually the result of the lack of papilla fill interdentally. With the improvement of dental procedures and materials, more attention has been directed to improving this unesthetic occurrence. Improvement of papilla loss (black triangle) can be mainly categorized into non-surgical and surgical techniques with most surgical modalities focused on a minimally invasive approach due to the restricted working area and blood supply to the papilla. Collagen matrix offers strong mechanical properties while promoting tissue healing and hence is used in many periodontal plastic surgeries (gum surgeries). However, the outcome of collagen matrix in treating papilla loss has not been studied yet. This study aimed to see at the clinical effects of collagen matrix in papilla augmentation using a minimally invasive surgical approach.

Patients with papillae loss were selected and Collagen matrix (Geistlich Fibro-Gide) used to stabilize the affected area with a minimally invasive surgical procedure. Papilla height gain, texture and color will be assessed pre-operatively, three and six months postoperatively. in addition, probing depth, clinical attachment level and keratinized tissue width will also be assessed.

DETAILED DESCRIPTION:
Introduction and Hypothesis of the Study:

The focus on achieving highly esthetic dental outcomes has increased nowadays, especially with the improvement of restorative and periodontal surgical techniques. Black triangles, an unesthetic occurrence due to lack of papilla, can occur when there is loss of the periodontal interproximal attachment apparatus. Plaque associated periodontal disease has been the most common reason for black triangle formation. However, it can also be caused by trauma, improper restorations contours, aggressive flossing, spacing between teeth and iatrogenic damage.

Patients with black triangles usually complain from unpleasant esthetic appearance, particularly when it harvests calculus, stains, and food. It usually gets worse with time requiring more attention in cleaning these open gingival embrasures using interdental brushes and floss.

Many surgical and non-surgical treatment modalities have been proposed as possible treatments for papilla loss. The non-surgical approach includes repeated root planning and curettage, and correcting contact points orthodontically to help induce papilla fill. Surgical papilla augmentation remains a challenge in periodontal regeneration due to the restricted interdental space and patterns of blood supply to the area. Many surgical techniques were suggested to overcome these challenges; semilunar incision where the papilla is left untouched, the use of a pedicle flap in a microsurgical technique without releasing incisions and papilla augmentation with customized connective tissue graft using the interproximal tunneling technique .The current literature on surgical correction techniques are mainly comprised of case reports and case series, and no standard surgical treatment of black triangles has been devised yet.

Collagen based matrices (CM) is a bovine-equine collagen-based tissue. Due to its strong mechanical properties, it acts as scaffold material for cell migration and helps in the overall healing process. CM has become very widely used and has proved its superiority in many periodontal procedures due to its excellent tissue color matching.

Due to the lack of clinical studies surrounding the use of collagen matrices in papilla augmentation, this study aims at investigating the effects of collagen matrices in papilla augmentation in patient with mild to moderate papilla loss. The primary objective of this study was to assess the papilla height gain in treated sites. The secondary objective was to compare the texture and color of the treated papilla to the respective patient's tissue. The hypothesis of this study was that CM will improve the papilla height gain and will look similar to the patient's periodontal tissue.

IV. Materials and Methods:

- Study Design and Ethical Considerations This study is a prospective clinical trial approved by the Internal Review Board (IRB) of Jordan University of Science and Technology before the commencement. Subjects were informed about the purposes and aims of the clinical procedure. The exact procedure along with possible complications were described to all patients. Patients were also informed about the advantages, safety and uses of collagen matrix material in soft tissue augmentations, particularly around dental implants. Patients were informed about other possible treatment options of black triangles.

Patients who agreed to be part of the study were assured of the confidentiality of all taken information and signed a written consent form. Participants were examined and full periodontal charting and scaling were done at least 2 weeks before the beginning of the treatment. Patients with periodontitis were referred to the periodontics clinic at Jordan University of Science and Technology. Participants were also advised to improve their oral hygiene practice before the beginning of the treatment.

Inclusion and Exclusion Criteria

- Inclusion Criteria

The fulfillment of inclusion criteria was verified during patients screening session. The included patients and sites to be treated met the following criteria:

* Male and female patients above the age of 18 years old with papilla loss.
* papilla loss between 2 natural teeth.
* Absence of active periodontal disease.
* Patients willing to follow oral hygiene measures.
* At least one papillary recession in the maxilla from UR5 to UL5.
* Papillay recession classified as 1 or 2 according to Nordland and Tarnow classification 1998.
* Sites with less than 7 mm measurement from the contact point to the bone crest.
* Sites having adequate width of attached gingiva(>2mm).

Exclusion Criteria

* Patients with incorrect crown or restoration margins, and/or caries.
* Patients undergoing orthodontic treatment.
* Patients who consume alchohol/smoking .
* Papilla loss around dental implant.
* Patients with any systemic disease that may compromise or affect the results of the surgical procedure.
* Breast feeding or pregnant woman.

Periodontal Examination

Full examination was conducted in the postgraduate periodontics clinic at The Dental Teaching Center in Jordan University of Science and Technology Using UNC-15 probe and sterile dental mirror. Measurements of pocket depth, O'leary plague index, bleeding on probing, clinical attachment loss were recorded on an examination sheet. The sheet also included the date and patient name. These measurements were taken to all participants to all facial sites extending from upper right second premolar to upper left second premolar as three readings for each tooth (mesial, mid facial, distal).

The distance from the contact point to the bone crest (transgingival probing), Interdental keratinized tissue width, papilla loss to nearest 0.5mm and Tarnow &Nordland classification were recorded for all papillary defect sites. In the present study, the above measures were taken at 3 points: baseline, 3 months, and 6 months.

All these measurements were taken as follows:

* pocket depth: the distance from the gingival margin to the sulcus depth.
* clinical attachment loss: the distance from cementoenamel junction to the sulcus depth.
* O'leary plaque index: recorded as 0 (no plaque on probing) or 1 (presence of plaque).
* bleeding on probing: recorded as 0 (no bleeding) or 1 (bleeding after site probing).
* bone sounding: the distance from the contact point to interdental bone crest.
* papilla loss reading: the distance from contact point to papilla tip to nearest 0.5 mm.

Sample Size

Patient screening and selection were conducted by a single, experienced postgraduate student in Periodontics. A sample of 30 sites was included in the present study. All participants included had at least 1 site with papilla loss between upper right to upper left second pre-molars. Sample size was calculated based on the change in the esthetic score.

Sample size calculation was performed using G power 3.1 software. The calculations were based on medium effect size (d = 0.5), an alpha level of 0.05, the desired power of 80%. The estimated sample size to detect a medium effect size in the change of esthetic score was 27 sites.

Selection of Cases Sites Case selection protocol involved a screening appointment to verify eligibility. Nearly all treated patients were seeking an esthetic solution for their papillary defects "black triangles". Some of them also expressed complaints of food impaction and phonetics air passages. All accepted cases had stable periodontal health, and a scaling visit was done at least two weeks before the surgery.

Surgical Procedure All patient signed a written consent form pre-surgically, which included procedure information, its purposes and possible complications.in addition to the dates of the reevaluation visits. Local anesthesia (articaine 0.4%) was administered facially at all papillary treated sites apically to the mucogingival junction, extended two teeth mesially and distally to the last treated papilla to allow for sufficient tunnelling laterally without causing any pain to the patient. Local anesthesia was also given palatal to the treated papilla sites.

Site Preparation In tunnel preparation, Intra-sulcular incisions with 15c blades were applied mesially and distally to the gingival slopes around interdental papillae. Care was taken to stay parallel to the teeth contour to avoid tearing the interdental papillae. intra-sulcular incisions in the middle gingival sites were made using tunnelling knife instead of the 15c blade to prevent any tearing to midfacial area.

All facial tissue was continuously tunneled with tunneling instruments apically to the mucoginigival line. All muscles and frenum attachments were detached internally though the tunnel by applying the tunneling knife parallel to the facial tissue. The separation of these attachments was completed with tactile sensation and at the end of this step, the facial tissues were easily moved coronally without any tension.

Interdental papillae were carefully reflected from the underlying crestal bone using the tunnelling knife in perpendicular direction if possible, or by using 11/12 Gracy curette. The curette was inserted through the tunnel facially and positioned over the interdental bone, then a coronal movement of the curette was applied until the point where interdental bone ended, and soft tissue began, felling it with tactile sensation. At this point, changing the direction of the curette while applying controlled force coronally was done to separate the interdental tissue from the underlying bone. This step was performed from the mesial and distal directions to all treated sites and the force was applied until interdental tissues could be freely moved towards the contact point.

The separation of the interdental tissue using Gracy curette. After performing this step on all treated sites, the facial and interdental tissue were freely moved coronally to the contact point area without any tension. Composite restorations were applied as interdental stops in the interproximal areas just coronal to the contact points avoiding any occlusal interferences. Etching was applied on mesial and distal line angles of the teeth and care taken not to reach the contact area with acid etch so that the restorations can be easily removed later.

Augmenting Fibro-Gide After preparation of papilla sites and the application of composite stops, 2 types of sutures were used. One to insert and fix the collagen matrix (Fibro-Gide®) and another to coronally advance the tissues. 4-0 nylon Suspension suture was used to coronally advance the tissue in each papilla site and 5-0 polyglycolic suture was used to insert and fix the collagen matrix (Fibro-Gide®) in each papilla site. First, nylon sutures were held in place without tightening to allow for the insertion of collagen matrix. Then, polyglactin suture (Vycril™) holding collagen matrix was inserted to reach the palatal tissue through the facially created tunnel.

Insertion of the collagen matrix was done though the sulcus, mesial or distal to the targeted papilla, by elevating the papilla gently and tucking the collagen matrix in though the created space.

Following securing the collagen matrix, polyglactin (Vycril™) and nylon sutures were fixed and secured to the composite stop. The same technique was then applied to the next papillary defect site until all collagen matrices were tucked and secured in the interdental tissue spaces.

In case of separation of the facial papilla from the palatal, additional 6-0 vicryl suture was applied from the tip of the separated papilla buccally to the tip of the palatal interdental tissue to ensure adequate primary closure over the augmented Fibro-Gide.

Post-Operative Instructions and Complication Management

Patients were instructed not to brush their teeth for 2 weeks and to rinse with chlorhexidine solution (0.2%) two times a day until the suture removal visit and to refrain from flossing or interdental brushing for 6 weeks. Patients were advised to use analgesics, such as nonsteroidal anti-inflammatory drugs on the first day. Subsequent doses were taken only if necessary. A soft cold diet was recommended for all patients particularly during the first days.

The sutures and composite restorations were removed at the two weeks' appointment. polishing was done to all upper and lower teeth. Interdental papilla sites were carefully examined, and the decision was made separately for each interproximal area regarding the use of an interdental toothbrush or dental floss at that site.

Parameters Assessed

Each site was evaluated individually. The following parameters were evaluated:

* Interdental Papilla Height (PAPILLA LOSS) Papilla loss was recorded presurgically, 3 and 6 months post-surgically using UNC-15periodontal probe by applying it parallel to the long-axis of the tooth. The reading was rounded to the nearest 0.5 mm. The amount of papilla loss was measured from the contact point to the tip of the papilla.
* Interdental Papilla Class Nordland and Tarnow classification system was used for each interdental papilla. The records were taken at baseline, 3 and 6 months post-surgically to detect any changes after the treatment.
* Normal: Interdental papilla fills embrasure space to the apical contact point/area.
* Class I: Tip of the interdental papilla lies between the interdental contact point and the most coronal extent of the interproximal cementoenamel junction.
* Class II: Tip of the interdental papilla lies at or apical to the interproximal CEJ but coronal to the apical extent of the facial cementoenamel junction.
* Class III: Tip of the interdental papilla lies level with or apical to the facial cementoenamel junction.
* Interdental Keratinized Tissue Width Keratinized tissue width was recorded to the nearest 1 mm from the tip of the papilla to the mucoginigival line. The record was taken using UNC-15 probe at baseline, 3 and 6 months.
* Digital Papilla Fill Papilla level measurements were taken digitally at baseline and 3 months. The distance from the contact point to the tip of the papilla was measured using measurement toll. To achieve this, the thirty treated papilla sites were recorded using intraoral optical scans (CEREC Omnicam, Dentsply Sirona). Then, all STL files were uploaded to exocad (DentalCAD 2.2 Valletta) software, and the measurements were taken using the measurements tool.
* Esthetic Score At three and six months, esthetic scores were recorded based on the esthetic score published by Cairo et al. (107). Each interdental papilla site received a score out of 10 depending on 5 variables: papilla level, papilla texture, papilla color, papilla contour and mucogingival alignment. Regarding the assessment of papilla level, 6 points was recorded if papilla was completely filled, 3 points if partial papilla fill occurred and 0 point if the level of the papilla stayed the same/got worse.

Whereas a score of 0 or 1 was used for each of the other variables:

* Interdental papilla texture: zero point = scar formation, papilla step present. 1 point= absence of a step/scar.
* Papillary color: zero point = color varies from adjacent/contralateral soft tissue. 1 point= normal healthy color that integrates with adjacent tissue.
* Papillary contour: zero point= improper papilla contour, flat. 1 point= proper scalloped contour.
* Mucogingival alignment: zero point= mucogingival junction not aligned with mucoginigival junction of adjacent teeth. 1 point= mucogingival junction aligned with mucoginigival junction of adjacent teeth.

Patient Centered Outcome Measures Each patient was given a questionnaire of 2 pages to evaluate pain attributes during the first 2 weeks. In addition, the overall esthetic satisfaction at baseline, three and six months post-operatively was recorded. The questionnaires were prepared based on the systematic review published by Stefanini and her coworkers.

Patients were asked to record a Visual Analog Scale (VAS) out of 10 for each of the following variables:

* Gingival and papilla Esthetic satisfaction pre-surgically, where 0 indicates no satisfaction and 10 indicates 100% satisfaction.
* Amount of stress pre-surgically, where 0 indicates no stress (peaceful) and 10 indicates very stressful.
* The degree of pain day 1 post-surgically, 0 indicates no pain, 10 indicates the most painful situation I have ever experienced.
* The degree of pain day 2 post-surgically, 0 indicates no pain, 10 indicates the most painful situation I have ever experienced.
* The degree of pain day 3 post-surgically, 0 indicates no pain, 10 indicates the most painful situation I have ever experienced.
* The degree of pain day 4 post-surgically, 0 indicates no pain, 10 indicates the most painful situation I have ever experienced.
* The degree of pain day 5 post-surgically, 0 indicates no pain, 10 indicates the most painful situation I have ever experienced.
* The degree of pain day (6-14) post-surgically, 0 indicates no pain, 10 indicates the painful situation I have ever experienced.
* Esthetic satisfaction at 3 months, 0 indicates no satisfaction and 10 indicates 100% satisfaction.
* Esthetic satisfaction at 6 months, 0 indicates no satisfaction and 10 indicates 100% satisfaction.
* The degree of esthetic improvement in comparison to baseline, 0 indicates no improvement,10 indicates very pleasant improvement.
* Overall results satisfaction, 0 indicates not satisfied, 5 indicates I am satisfied but I would not do the surgery again and 10 indicates I'm satisfied and ready to do the surgery again.
* Did the treatment improve your quality of life? 0 indicates no improvement, 10 indicates very large improvement.

Additionally, the questionnaire included the following yes or no questions:

Did bruising occur? Swelling on day 0? Swelling on day 1? Swelling on day 2? Swelling on day 3? Swelling on day 4? Swelling on day 5? Swelling from days 6-14?

ELIGIBILITY:
Inclusion Criteria

* Male and female patients above the age of 18 years old with papilla loss.
* papilla loss between 2 natural teeth.
* Absence of active periodontal disease.
* Patients willing to follow oral hygiene measures.
* At least one papillary recession in the maxilla from UR5 to UL5.
* Papillay recession classified as 1 or 2 according to Nordland and Tarnow classification 1998.
* Sites with less than 7 mm measurement from the contact point to the bone crest.
* Sites having adequate width of attached gingiva(>2mm).

Exclusion Criteria

* Patients with incorrect crown or restoration margins, and/or caries.
* Patients undergoing orthodontic treatment.
* Patients who consume alchohol/smoking .
* Papilla loss around dental implant.
* Patients with any systemic disease that may compromise or affect the results of the surgical procedure.
* Breast feeding or pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
papilla height | 6 months
  papilla loss , papilla height reduction , before and after the surgery measuring from contact point to interdental tissue level.

SECONDARY OUTCOMES:
esthetic score, texture,color,contour | 6 months
  esthetic score at 3,6 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: dr reem sami abdelhafez prof rola alhabashneh, prof, Study Director — Jordan University of Science and Technology; Bahaaaldin Alsharif, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan